CLINICAL TRIAL: NCT02531243
Title: A Pilot Study of Computerized Biofeedback Games With Young People Experiencing Psychotic-Spectrum Symptoms
Brief Title: Computer-Aided Learning for Managing Stress
Acronym: CALMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kristen Woodberry, Director, Program for Psychosocial Protective Mechanisms, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000377; K23MH102358 (NIH)
Record Dates: First submitted 2015-07-13; First posted 2015-08-24 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Psychosis
Keywords: prodrome; family therapy; clinical high risk
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CALMS (Experimental): 12 session family therapy using multi-user biofeedback games
  Interventions: Behavioral: CALMS

INTERVENTIONS:
Behavioral: CALMS — Family Therapy; Multi-user Biofeedback Videogames

SUMMARY:
The purpose of this study is to learn whether a new family therapy using computer games with biofeedback might help people at clinical high risk for psychosis and their family members learn to experience less stress and have fewer mental health challenges.

DETAILED DESCRIPTION:
CALMS revolves around the use of Emotional Manipulatives (EM) developed at Boston Children's Hospital (BCH). EM are single and multi-user biofeedback games designed to enhance executive control of emotion. The intervention and EM in CALMS were adapted from those used in Anger Control Training (ACT) with Regulate and Gain Emotional Control (RAGE-Control). In a randomized controlled trial at BCH, ACT and RAGE-Control relative to "sham" video-game play without biofeedback led to significantly greater reductions of aggression in adolescents and greater improvement in family functioning.

In this feasibility study, family dyads will participate in 12 sessions aimed at

1. enhancing engagement through the use of video and other games,
2. enhancing stress resilience through biofeedback, education, and individualized stress-reduction practice, and
3. harnessing the power of the family to enhance contextual learning and the generality and duration of effects.

Clinical, self-report, and heart rate measures will be assessed at baseline, 4, 8, and 12 week assessments.

ELIGIBILITY:
Inclusion Criteria:

* Currently Meet or Have Met Criteria of Prodromal Syndromes (COPS) according to the SIPS within the past 2 years
* Estimated IQ > 70
* Speak fluent English
* Have at least one parent or adult family member who also speaks fluent English and is willing to participate

Exclusion Criteria:

* Physical limitations precluding effective use of biofeedback videogames
* Co-morbid psychiatric disorders, including substance disorders, but only if they better explain COPS symptoms or make participation counter-indicated.
* Active suicidal ideation or attempts within the past 2 months unless being actively monitored and treated for this by a clinician

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Feasibility: Percent of referred who consent and meet study criteria | Up to six months
  Enrollment
Feasibility: Percent of 12 sessions completed | Up to six months
  Engagement: Percent of sessions completed by consented and eligible participants
Feasibility: Counts of premature termination of intervention | Up to six months
Feasibility: Self-report of Credibility/Satisfaction | 12 week assessment or last assessment completed
  Individual and family member self-report
Feasibility: Self-report of User Experience | 12 week assessment or last assessment completed
  Self-report of ability to learn/use technology to lower stress reactivity

SECONDARY OUTCOMES:
Change in Perceived Stress relative to Baseline | Weeks 4, 8, and 12 Assessments
  Self-report via Perceived Stress Scale
Change relative to Baseline in Youth Perceptions of Relationship with Family Member | Weeks 4, 8, 12 Assessments
  Self-report of conflict, criticism, and warmth in relationship with participating family member
Change relative to Baseline in Parent Perceptions of Relationship with Adolescent or Young Adult | Weeks 4, 8, 12 Assessments
  Self-report of conflict, criticism, and warmth in relationship with youth
Positive Symptom Score Change relative to Baseline | Weeks 4,8, and 12 Assessments
  Total positive symptom score according to the Structured Interview of Psychosis-risk Syndromes (SIPS)
Change in Social and Role Functioning relative to Baseline | Weeks 4, 8, and 12 Assessments
  Global Functioning: Social & Role Scales;
Change in Global Functioning relative to Baseline | Weeks 4, 8, and 12 Assessments
  SIPS Global Assessment of Functioning
Safety: Change in Hostility/Aggression relative to Baseline | Weeks 4, 8, and 12
  Self-report
Safety: Change in Video-game Addiction relative to Baseline | Weeks 4, 8, and 12
  Self-report
Difference in reaction times for emotional and calm faces on an Emotional Go/NoGo Task | Baseline, Weeks 4,8, and 12
  Executive Control of Emotion

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Woodberry, MSW, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodberry KA, Chokran C, Johnson KA, Nuechterlein KH, Miklowitz DJ, Faraone SV, Seidman LJ. Computer-aided learning for managing stress: A feasibility trial with clinical high risk adolescents and young adults. Early Interv Psychiatry. 2021 Jun;15(3):471-479. doi: 10.1111/eip.12958. Epub 2020 Apr 1. PMID 32237208